CLINICAL TRIAL: NCT01936662
Title: Endotracheal Intubation vs. Laryngeal Mask Airway for Esophagogastroduodenoscopy in Children
Brief Title: Endotracheal Tube Versus Laryngeal Mask Airway for Esophagogastroduodenoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1011002885
Record Dates: First submitted 2013-08-29; First posted 2013-09-06 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Airway Morbidity
Keywords: Airway management comparison

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Largyngeal Mask Airway for EGD procedure (Experimental): Patients randomized to LMA to maintain airway through EGD procedure
  Interventions: Device: LMA
- Endotracheal Tube for EGD procedure (Active Comparator): Patients were randomized to ETT to maintain airway for EGD procedure. This is the standard of care at this hospital
  Interventions: Device: ETT

INTERVENTIONS:
Device: LMA — Patients randomized to the LMA group had their airways maintained with a LMA device
  Arms: Largyngeal Mask Airway for EGD procedure
Device: ETT — Patients assigned to this group had an ETT placed to maintain their airway, as is standard of care at this hospital
  Arms: Endotracheal Tube for EGD procedure

SUMMARY:
Esophagogastroduodenoscopy (EGD) is a relatively common procedure in pediatric patients undergoing evaluation for various gastrointestinal ailments. The procedure itself, with or without associated biopsies, is relatively short in length. Unlike adults, who regularly undergo this procedure with conscious sedation, children most often require general anesthesia. While safe and effective, endotracheal tracheal tube (ETT) intubation of children for EGD can result in delayed awakening and slow room turnover, particularly when intravenous medications are required for intubation. Laryngeal mask airway (LMA) is an alternative to intubation, which permits removal before full awakening.

Although considered a safe alternative to tracheal intubation in appropriate cases, disadvantages of the LMA have been reported including kinking, occluding view of the surgical field, failure of placement requiring tracheal intubation, aspiration of gastric contents, desaturation, and laryngospasm. The study was designed to determine whether use of an LMA for EGD could reduce operating room time, while providing satisfactory conditions for the endoscopist, and an equivalent side effect and safety profile as compared to ETT in otherwise healthy children with gastrointestinal complaints

DETAILED DESCRIPTION:
1. Study design The study will be randomized, controlled, and prospective in design.
2. Comparison groups The two comparison groups will be:

   1. Laryngeal Mask Airway Group (LMA), N = 42 LMA will be used as the intraoperative airway device.
   2. Endotracheal Tube Group (ETT), N = 42 ETT will be used as the intraoperative airway device.
3. Study and timeline of interventions

   1. Preoperative: All patients enrolled in this study will receive a standard preoperative dose of oral midazolam 0.5 mg/kg up to 15 mg, 15 to 30 minutes prior to anesthetic induction.
   2. Intraoperative: Subjects will all undergo induction of anesthesia by inhalation of sevoflurane and oxygen. An intravenous catheter (IV) will be placed, followed by lidocaine 2mg/kg IV. The airway device will be placed (LMA or ETT). As required for the procedure, the subject will be placed in a left lateral decubitus (left side down) position. Maintenance of anesthesia will be provided with sevoflurane at a concentration of 1.5-2 MAC, or higher if deemed appropriate for the clinical setting as judged by the anesthesiologist. All participants will be given the anti-nausea medicine ondansetron 0.1mg/kg (maximum 4 mg) after placement of the airway device. When the endoscope is removed at the completion of the procedure, the patient will be returned to the supine position. The sevoflurane will be discontinued and the airway device will be removed when the anesthesiologist deems it appropriate. Prior to leaving the OR, the anesthesiologist may give pain or anti-anxiety medicine as needed.
   3. Postoperative: All patients will receive routine PACU care. Pain and anxiety scores will be recorded according to routine PACU practice. Medication for pain, nausea, and anxiety will be given according to the judgment of the anesthesiologist.
   4. Measured end-points:

   i. Time from induction of anesthesia to placement of the airway device ii. Time from end of procedure to arrival in the PACU iii. Time spent in the PACU iv. Overall time from arrival in the OR to discharge home v. Vomiting after the procedure vi. Nausea requiring medicine after the procedure vii. Lowest oxygen saturation level during or after the procedure viii. Highest concentration of sevoflurane during the procedure ix. Highest pain level after the procedure x. Amount of pain medicine given xi. Adverse events xii. Satisfaction level of the doctor doing the EGD

ELIGIBILITY:
Inclusion Criteria:• Age 3-17

* Scheduled for Esophagogastroduodenoscopy, with or without biopsies
* Have been informed of the nature of the study and informed consent has been obtained from the legally responsible
* Have provided assent in accordance with Institutional Review Board requirements
* Are able to complete pain assessment evaluations as determined by preoperative evaluations

Exclusion Criteria:

* • Abnormal/difficult airway

  * Symptomatic obstructive sleep apnea
  * Risk of aspiration of stomach contents
  * Upper respiratory infection within last 14 days
  * Allergy to lidocaine or ondansetron
  * EGD procedures associated with the need to exclude ondansetron administration
  * BMI >85th percentile for age
  * Are unable to communicate effectively with study personnel
  * Have a positive urine pregnancy test (menstruating females only at screening

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micahel Acquaviva, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Acquaviva MA, Horn ND, Gupta SK. Endotracheal intubation versus laryngeal mask airway for esophagogastroduodenoscopy in children. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):54-6. doi: 10.1097/MPG.0000000000000348. PMID 24637966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited on the day of their scheduled endoscopic procedure in the outpatient clinic of a large children's hospital.
Pre-assignment Details: Patients were pre-screened for allergies to medications used and BMI's outside the 90th percentile. All other patients were eligible for enrollment.
Groups:
- LMA Used to Maintain Airway: Patients randomized to LMA to maintain airway through EGD procedure
- ETT Used to Maintain Airway: Patients were randomized to ETT to maintain airway for EGD procedure. This is the standard of care at this hospital
Period: Overall Study
Arm/Group | LMA Used to Maintain Airway | ETT Used to Maintain Airway
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMA Used to Maintain Airway | ETT Used to Maintain Airway | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 42 | 84
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (6.2) | 10.1 (4.2) | 10.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Endoscopist Satisfaction
Description: Endoscopist was surveyed to determine their satisfaction with each of the airway devices.
  Endoscopist used the following satisfaction scale for each patient, regardless of the airway device used:
  1. The airway device did not interfere at all with the ability to perform the scope.
  2. The airway device presented some interference with the scope, but not enough to cause difficulty.
  3. The airway device made it difficult to perform the endoscopy.
  4. The airway device prevented the endoscopy from being performed.
Time Frame: 2 hours
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Largyngeal Mask Airway for EGD Procedure | Endotracheal Tube for EGD Procedure
Number analyzed (Participants) | 42 | 42
units on a scale | 1.0 (0.0) | 1.1 (0.3)

2. Secondary Outcome: OR to Discharge (Min)
Description: Overall time from arrival in the OR to discharge home (in minutes)
Time Frame: OR to discharge
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | LMA Used to Maintain Airway | ETT Used to Maintain Airway
Number analyzed (Participants) | 42 | 42
Minutes | 86.6 (18.5) | 102.5 (40.4)

ADVERSE EVENTS:
Arm/Group | LMA Used to Maintain Airway | ETT Used to Maintain Airway
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LMA Used to Maintain Airway (N=42) | ETT Used to Maintain Airway (N=42)
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
asthma exacerbation postop (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes